CLINICAL TRIAL: NCT06938048
Title: Effectiveness of Short-stretch Bandages for Treatment of Hand Edema Compared to High Stretch Bandage: Cross Over Randomized Controlled Trial (RCT)
Brief Title: COMPARISON OF BANDAGE IN HAND EDEMA
Acronym: Hand bandage
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Regione del Veneto - AULSS n. 7 Pedemontana (Other)
Responsible Party: Principal Investigator, Silvia Fontana, Medical Doctor, specialized in Physical Medicine and Rehabilitation, head of Hub Lymphedema Center AULSS 7 Pedemontana, Regione del Veneto - AULSS n. 7 Pedemontana
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 280CET
Record Dates: First submitted 2025-01-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-01

CONDITIONS: Edema
Keywords: bandages; edema; hand
MeSH Terms: conditions — Edema | interventions — Monensin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm "Short First" (Experimental): Short stretch bandage applied in the first 24 hours
  Interventions: Other: short stretch bendage (Lohmann e Raucher); Other: high stretch bandage (Coban)
- Arm "High first" (Active Comparator): High stretch bandage applied in the first 24 hours
  Interventions: Other: short stretch bendage (Lohmann e Raucher); Other: high stretch bandage (Coban)

INTERVENTIONS:
Other: short stretch bendage (Lohmann e Raucher) — extensibility between 10% to 100% of the lenght
Other: high stretch bandage (Coban) — extensibility above 100% of the lenght

SUMMARY:
The aim of this clinical trial is to compare the effectiveness of high and short stretch bandages in hand edema treatment of adult patients with affected hand volume superior of at least 5% compared to the contralateral hand. The main question to be answered by this study is: which bandage is more effective in reducing edema?

Endpoint 1: hand volume, measured by immersion volumetry (Valgrado method). Endpoint 2: ROM (range of motion) of the fingers and wrist, measured by goniometry.

Endpoint 3: Results of a semi-structured interview on participants subjective perception of hand function and esthetics, ADL performance and quality of life.

This study includes 2 groups (arms); each participantreceives both types of bandages but in a different temporal order depending on group membership:

* Arm A: short stretch bandage applied as the first treatment.
* Arm B: high stretch bandage applied as first treatment. Patients will be randomized 1:1 using the RedCap Software.

The entire study will take place over 3 consecutive days. On each of these days, participants are examined (hand volume, finger and wrist ROM), receive the bandage (the type of bandage depends on the participant group), undergo physiotherapy treatment and then practice specific hand mobilization exercises at home.

At the end of the study, the data on hand volume and mobility of the hand and wrist will be analyzed to determine which type of bandage, high-stretch or low-stretch one, is most effective in reducing hand volume (and therefore hand edema) and mobility of the hand and wrist.

In addition, data collected using the semi-structured interview will be analyzed to examine patients subjective perceptions of hand function and esthetics, ADL performance and quality of life.

DETAILED DESCRIPTION:
Aims of the study

This study has one primary aim and two secondary aims. The primary aim is to find out which bandage is more effective in the treatment of hand edema in orthopaedic patients. The short-stretch bandage will be compared with the high-stretch bandage, with the latter being more commonly used. The effectiveness of the bandage in the treatment of hand edema is demonstrated by its ability to reduce the volume of the affected hand. The first secondary objective is to investigate the patients' subjective perception regarding the impact that hand edema and the application of the bandage may have on the function and aesthetic appearance of the hand, performance of ADLs and quality of life. The study is carried out by giving the participating patients a specific semi-structured interview. The second secondary objective is to measure the passive joint ROM of the wrist and the five fingers of the hand: metacarpophalangeal, proximal interphalangeal, distal interphalangeal. This is performed to assess any improvement in passive joint ROM between before and after application of the bandages, which should follow the reduction in hand edema caused by the bandages. The "conical" shape of the finger is well suited to evaluate the effectiveness of a bandage. If the tension of the bandages is the same, distal pressure is greater than the proximal pressure (Laplace's law: the pressure is inversely proportional to the radius of curvature and proportional to the tension). This reduces the possibility of error errors caused by incorrect application of the bandage. In addition, the movement of the fingers and hand, required for the patients in the study by performing specific exercise program at home, in addition to promoting pressure peaks that favor fluid advancement, allows normalization of the tension of the coils of the bandage.

Study design

The identified study design is a randomized, controlled trial with cross-over (RCT with cross-over). The study is multicenter and has no commercial purpose (no profit). Patients with hand edema who meet the inclusion and exclusion criteria, will be included and then randomized into the two study groups.

Randomization

Patients in this study will be randomized in a 1:1 ratio, by simple randomization, into the following two groups: Group A - experimental (short-stretch bandage for the first 24 hours, high-stretch bandage for the next 24 hours); Group B - control (high-stretch bandage for the first 24 hours, short-stretch bandage for the next 24 hours).

The randomization procedure is performed with the REDCap platform.

Cross-over

This study is a a cross-over as each patient receives both types of bandages, regardless of the group to which they belong. The cross-over makes it possible to reduce the sample size, and still obtain statistically significant results. The only thing that changes between the experimental group and the control group, is the timing of the application of the two different types of bandage: the materials used, the procedures and the assessments performed are the same in both groups.

Study blinding

This study is blinded because the patient and the outcome assessor are blinded to the type of bandage used (high or short stretch) and therefore the group to which the patient belongs (experimental or control). The patient does not know what type of bandage is being applied, as the physiotherapist applying the bandage does not tell the patient what type of bandage is being used. The endpoint evaluator also does not know what type of bandage the patient is wearing, as he is not present when the patient is bandaged and performs his assessment with the patient's unattached hand. In fact, each patient in the study is explicitly instructed by their physiotherapist to remove the bandage on their own approximately 30 minutes before the examination. In addition, both the patient and the endpoint evaluator are kept separate from the randomization process and the patient group (Group A or B).

Study setting

This study is multicenter and the participating centers are:

* UOC of Functional Recovery and Rehabilitation of the Alto Vicentino Hospital.
* Professional clinic "Elena Lanfranchi".
* Fisiomed Polyclinic.

Endpoints of the study

1. Volume of the edematous hand, measured by Valgrado volumetry.
2. Passive ROM (range of motion) of the wrists and the five fingers of the edematous hand (metacarpophalangeal and interphalangeal joints).
3. Scores of the different areas assessed by the semi-structured interview.

Variables of the study

The dependent variables correspond to the endpoints listed above. The independent variable is represented by the type of hand bandage applied.

Protective factors

The protective factors are represented by:

* The person performing the treatments is different from the person performing the assessment.
* The person carrying out the examination does not know what kind of bandage the patient is wearing.
* The patient himself does not know what type of bandage he was wearing.
* The bandages are applied in the same way in both groups of the study (experimental and control group).

Risk factors

Each unit in the sample receives two different bandages, one after the other, without a time break in between. A possible risk factor is that the first dressing applied may cause a greater reduction in hand volume than the second dressing applied (which is applied to a hand that has already experienced a reduction in edema from the previous dressing).

No washout in the study

The time-dependent reduction in pressure exerted by short-stretch bandages is a well-known phenomenon and is related to the decrease in volume of the bandaged body part and the partial relaxation of the bandages. (Damstra R.J., Brouwer E.R. et al.) This significant and rapid drop in pressure with short-stretch bandages means that the bandage must be replaced daily in the initial phase of compression therapy. (Todd M.) This information justifies the lack of need to allow a certain amount of time to elapse between the application of the two bandages in the present study (wash-out). By the time the second bandage is applied, the first bandage has already had its effect and can be considered ineffective. We also consider this reasonable because the pressure exerted by short-stretch bandages is already reduced by 1/3 30 minutes after application, as mentioned in this study (Damstra R.J., Brouwer E.R. et al). The main reason for this rapid reduction in the pressure exerted by short-stretch bandages is the (therapeutic and intentional) reduction in the volume of the bandaged body part, which is achieved immediately after application of the bandage in both lymphoedema- affected and healthy subjects.

Bias

* The treatments (bandages) are performed by different people. This bias was eliminated because the methods for applying the bandages were exchanged before the start of the study and all experimenters underwent practical training. In addition, an explanatory video on the correct method of dressing application was produced and distributed to all experimenters.
* Presence of patients with edema of different origin (traumatic or surgical), in the acute phase (within 6 months of trauma). However, the literature studies show a similar heterogeneity of the sample with edema of different etiologies. In addition, edema is classified not so much by etiology, but rather by whether it is acute (within 6 months of onset) or chronic (more than 6 months after onset).

  * Selection bias: the differences found between the experimental and control groups are reduced by carrying out a randomized, controlled, cross-over study.
  * Measurement bias: the different centers participating in the study use different measurement instruments but meeting the same standards. In particular, the scale used is a high-resolution and high-capacity scale: resolution of 1 g and capacity of 6 kg. The brand of the instrument may vary but not its characteristics, which are standardized among the different centers participating in the study.
  * Performance bias: The patient and the endpoint evaluator are blind to the type of bandage the patient receives. The investigator, on the other hand, knows which bandage is used because he applies it himself.

DATA COLLECTION TOOLS

Exercises suggested to the patients in the study

Considering the data in the literature, it is clear that the positive effects of active exercise on edema cannot be overlooked and that active exercise must be an integral part of treatment. In fact, each patient in the present study will be educated and trained in the correct execution of three active mobilization exercises for the bandaged hand to be performed at home while wearing the bandage. The three exercises in question are selected by the patient's physiotherapist from the exercises listed in the exercise program developed for this study. These three exercises are those that are most appropriate based on the patient's clinical characteristics. During the 24 hours in which the first bandage is applied and during the 24 hours in which the second bandage is applied, each patient performs the same 3 exercises chosen for him by his physiotherapist, regardless of the type of bandage, and at the same dosage. Therefore, the dosage to be respected by the patients when performing the exercises is the same on the different days of the study and is the same for all patients: 10 repetitions for each exercise, performing all the selected exercises at least 3 times per day, as suggested by (Mackin E.J.). To encourage compliance with the treatment and correct execution of the exercises, each patient receives a booklet with illustrations of the proposed exercises. This booklet was created by the experimenter specifically for this study and contains exercises that involve active mobilization of all joints of the fingers and hand as suggested by (LaStayo P., Winter K. et al) and (Skirven T.M., Osterman A.L. et al). In the booklet, each exercise is described in simple terms and accompanied by a photograph on the side demonstrating its execution.

Finally, for each patient in the study, the performance of the exercises at home is examined during the semi-structured interview, which includes specific questions on this topic.

Valgrado volumetry

Valgrado volumetry is a technique for measuring hand volume that uses Archimedes' principle and takes less time than the classic volumetric method. In Valgrado volumetry, the hand is immersed in a vessel filled with water (not to the brim), which is placed on a precision scale connected to a PC that processes the data directly. This instrument minimizes measurement errors due to limb movements. The instrument used in the present study is a core balance with a capacity of 6 kg and a sensitivity of 1 gram. The results of this study (Hughes S., Lau J.) suggest that Valgrado volumetry has the same accuracy and precision as the classical volumetric method, and even has the potential to provide more accurate and precise results.

In addition, Valgrado volumetry is faster than the classical volumetric method: a single measurement of hand volume with the classical volumetric method takes about 45 seconds (Pellachia G.), while with Valgrado volumetry it takes about 16 seconds. Consequently, this latter technique offers the possibility of increasing the number of volumetric measurements that can be performed in the same session, thus increasing the statistical value of the assessment. Before performing volumetry, the hand to be examined must first be properly washed and dried, and the limit of immersion in water must be determined. The hand to be examined is then immersed in water up to this limit, taking care not to touch the bottom and sides of the container.

In the present study, the boundary of hand immersion in water is identified as the imaginary line connecting the spinous processes of the radius and ulna. The following procedure is used to locate this line. The patient sits on a chair, hand and forearm are pronated and rest on a table. The examiner places his index finger and thumb near the spinous processes of the radius and ulna on the dorsal side of the patient's wrist. The examiner then places a ruler on the dorsal surface of the patient's wrist, distal to but in contact with his fingers, and then releases his hand (whose thumb and index finger were positioned in line with the spinous processes of the radius and ulna), but keeps the ruler in the previously identified position. Next, the examiner stabilizes the patient's hand in the volumeter in the desired position for evaluation (i.e. with the meniscus of the water of the volumeter in line with the previously identified line on the patient's wrist). To do this, the examiner supports and stabilizes the patient's forearm with his own hands, taking care not to touch the bottom and sides of the container with the patient's hand and not to insert his own hands into the water. While the examiner stabilizes and supports the patient's forearm as described, he sits on a stool directly next to the patient and supports his own elbows against his own thighs. This allows the examiner to better stabilize the patient's hand in the desired position, reduce the oscillations of the volumeter's water and thus increase the statistical quality of the measurement.

Measurement of wrist and fingers ROM

Measurement of the ROM of the wrist and fingers is essential for a correct and complete physical examination of the hand. (Lane J.G., Gobbi A.) Since persistent edema has a direct negative impact on joint range of motion (ROM) and the purpose of this study is to determine which brace is most effective in treating hand edema, this study includes, among other things, measurement of passive joint ROM of the wrist and five fingers of the hand (metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints). This is done to assess any improvements in passive joint ROM before and after application of the supports, which should result from the reduction in hand edema caused by the supports. The degrees of freedom assessed for each of the joints mentioned are flexion and extension. The measurement is performed with a special finger goniometer.

Semi-Structured Interview

As part of the present study, a semi-structured interview was administered to each participant. This interview was specifically developed by the experimenter for the purposes of this research, with the aim of exploring patients' subjective perceptions regarding the impact of hand edema and the applied bandage on hand function, aesthetic appearance, performance of activities of daily living (ADLs), and overall quality of life.

The design of the interview was based directly on findings from a comprehensive review of the scientific literature. It investigates not only the main reasons for non-adherence to or discontinuation of compression therapy, but also patients' subjective experiences and perceived quality of life during treatment with compression bandages.

The response options used in the interview mirror those of the validated Italian version of the Lymphedema Quality of Life Questionnaire (LYMQOL) (Monticone M., Ferriero G. et al.). Additionally, some of the interview questions were adapted from existing questionnaires in the literature that assess quality of life and the impact of edema on individuals affected by the condition. Finally, as previously described, the study requires each participant to perform three active mobilization exercises of the bandaged hand at home. To assess the execution of these exercises, the semi-structured interview includes specific questions addressing this aspect.

The interview is administered to each patient at two separate time points:

First administration: after the removal of the first bandage and before the application of the second one; Second administration: after the removal of the second bandage. During each administration, the questions related to the bandage specifically refer to the one worn in the previous 24 hours. This is clearly explained to each patient prior to the interview.

Bandage Application Method

Both types of bandages examined in this study (short-stretch and high-stretch) are applied using the same standardized method, described as follows. The bandage is first secured with a loop around the wrist, proceeding from the radial side (radial styloid process, dorsal aspect) to the ulnar side (ulnar styloid process, dorsal aspect), with the hand and forearm in a pronated position. It is then passed over the back of the hand toward the distal phalanx of the fifth finger.

The bandage is applied in a circular manner around the finger, placing a single layer that overlaps the previous layer by two-thirds. The nail surface is intentionally left uncovered. Once the metacarpophalangeal joint of the fifth finger is reached, the bandage is passed again over the back of the hand, around the wrist, and then directed toward the fourth finger. Each finger, from the fourth to the first, is bandaged using the same method as for the fifth, always anchoring the bandage at the wrist before moving to the next finger. The palm is left unbandaged, while the dorsal surface of the hand is completely covered. During application, the bandage roll must remain in contact with the skin at all times. The bandage should not be stretched, but rather gently wrapped around the hand, using only the natural tension generated by the rolling motion. Once the first roll is finished, a second roll is applied starting from the wrist, following the same procedure.

Prior to the start of the study, the bandage application method was standardized and shared among all experimenters, who also received hands-on training. Additionally, an instructional video demonstrating the correct application technique was created and distributed to all experimenters.

Study Procedures

The study is conducted over three consecutive days. During this period, each participant-regardless of their assigned group-undergoes the same standardized set of procedures, as detailed below:

Day 1 of Treatment (T0)

The patient undergoes the first physiotherapy session, which consists of the following steps:

1. Assessment: Measurement of hand volume and joint range of motion (ROM) of the wrist, as well as the metacarpophalangeal and interphalangeal joints of all five fingers, using the tools and methods previously described.
2. Therapeutic exercises and rehabilitation treatment.
3. Application of the first bandage: The type of bandage applied depends on the patient's group allocation (Group A - experimental: short-stretch bandage; Group B - control: high-stretch bandage).
4. Patient education and training: Instruction in the correct performance of three active hand mobilization exercises to be carried out at home while wearing the bandage. The physiotherapist selects the three most appropriate exercises for the individual patient from the standardized exercise program.
5. Instruction on bandage removal: The physiotherapist explains how to correctly remove the bandage independently. The patient is instructed to remove the bandage 30 minutes prior to the second physiotherapy session, scheduled for the following day.

Day 2 of Treatment (T1)

The patient undergoes the second physiotherapy session, which includes:

1. Removal of the first bandage: In accordance with prior instructions, the patient independently removes the bandage 30 minutes before the session.
2. Assessment: Re-evaluation of hand volume and joint ROM of the wrist and fingers, conducted as on Day 1.
3. Administration of the semi-structured interview: The interview focuses on the patient's experience with the first bandage.
4. Therapeutic exercises and rehabilitation treatment.
5. Application of the second bandage: The type of bandage applied is based on the group allocation (Group A - experimental: high-stretch bandage; Group B - control: short-stretch bandage).
6. Review of home exercises: The three active mobilization exercises previously selected are reviewed with the patient.
7. Reinforcement of bandage removal instructions: As on the previous day, the patient is instructed to independently remove the bandage 30 minutes before the third physiotherapy session.

Day 3 of Treatment (T2)

The patient attends the third physiotherapy session, which includes:

1. Removal of the second bandage: As previously instructed, the patient independently removes the bandage 30 minutes prior to the session.
2. Assessment: Measurement of hand volume and joint ROM, performed using the same procedures as on the previous days.
3. Administration of the semi-structured interview: This interview focuses on the second bandage.
4. Therapeutic exercises and rehabilitation treatment.
5. Application of a hand bandage: The final bandage applied at the end of the third session is selected at the discretion of the treating physiotherapist, based on clinical judgment. This bandage is not part of the study protocol.

Follow-Up Follow-up assessments are conducted at 24 hours (T1) and 48 hours (T2). Each bandage is worn for a period of 24 hours, and patients are reassessed at the time of its removal.

ELIGIBILITY:
Study Population A total of 45 patients will be recruited for this study, according to the following inclusion and exclusion criteria.

Inclusion Criteria

* Presence of hand edema, with the affected hand showing a volume at least 5% greater than the contralateral hand. Hand volume is measured using the Valgrado immersion volumetry method.
* Edema of the following etiologies:

  * Traumatic (injury to the hand or upper limb resulting in edema of the hand or fingers)
  * Surgical
  * Algodystrophic
  * Rheumatologic
  * Secondary to immobility

Exclusion Criteria

* Lacerations or cut injuries to the forearm, due to the potential compromise of lymphatic drainage pathways from the hand.
* Edema of etiologies other than those specified in the inclusion criteria. Specifically, edema due to infection or structural and/or functional impairment of the lymphatic system-of any nature, including iatrogenic-is excluded.
* Pathologies involving the peripheral nervous system of the upper limb (e.g., nerve injuries with resulting paralysis).
* Contraindications to active mobilization of the wrist and finger joints (metacarpophalangeal and interphalangeal joints).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hand volume | Hand volume will be measured 3 times, from enrollment to 48 hours after: T0 (first assessment), T1 (24 hours after first bandage application), T2 (24 hours after second bandage application).
  Hand volume will be measured using immersion volumetry, according to the Valgrado method.

SECONDARY OUTCOMES:
Range Of Motion (ROM) | Wrist and fingers ROM will be measured 3 times, from enrollment to 48 hours after: T0 (first assessment), T1 (24 hours after first bandage application), T2 (24 hours after second bandage application).
  ROM of the wrist and hand joints-including the metacarpophalangeal and interphalangeal joints of all five fingers-will be assessed using standard goniometry.
Semi-structured interview | Results from the semi-structured interview will be collected 2 times, from enrollment to 48 hours after: T1 (24 hours after first bandage application), T2 (24 hours after second bandage application).
  Data on each participant's subjective perception of hand function and aesthetics, performance of activities of daily living (ADLs), and quality of life will be collected using a semi-structured interview specifically developed for this study.

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS 7 Pedemontana, Bassano, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
IPD must be submitted to local Ethical Committee